CLINICAL TRIAL: NCT02443818
Title: Non-randomised Open Label Pilot Study of Sirolimus Therapy for Segmental Overgrowth Due to PIK3CA- Related Overgrowth
Brief Title: Sirolimus Effect on Hypertrophic Syndromes Related Gene PIK3CA
Acronym: PROMISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLIVIER-FAIVRE Sirolimus
Record Dates: First submitted 2015-05-04; First posted 2015-05-14 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Segmental Overgrowth Disorders Due to PIK3CA
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Low dose sirolimus will be given in daily dosing to achieve trough levels of 2-6 ng/ ml.

SUMMARY:
It was found that people who have an excessive growth in one or more parts of their body and normal growth in other parts, may have a change in genes responsible for controlling cell growth. This genetic discovery identified a possible treatment for this overgrowth, called Sirolimus.

This is a pilot study, which help the investigators prepare a larger international study, which will aim to determine whether a treatment based Sirolimus is able to stop the excessive growth of one or more parties of their body in people who carry a genetic change in the PIK3CA gene (phosphatidylinosilol-3-kinase encoded by the gene PIK3CA).

DETAILED DESCRIPTION:
The duration of participation is 15 months:

* Visit screening: blood test, pre-clinical evaluation, urine collection and chest X-ray.
* First 6 months: participants will have their overgrowth monitored. This step includes 2 visits taking place at the University Hospital of Dijon: complete clinical evaluation, MRI of the body part by the overgrowth and Dual-energy X-ray absorptiometry (DXA).
* Next 6 months: participants will take Sirolimus. This step includes 2 visits (4 and 13 weeks after the start of treatment at local hospital): blood test, urine collection and clinical evaluation.

and 1 end of study visit after 6 months of treatment taking place at the University Hospital of Dijon: blood test, complete clinical evaluation, urine collection, MRI and DXA.

Participants will have several blood and urine tests between visits (1 and 2 weeks after the start of treatment at a local laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Post-zygotic PIK3CA mutation
* Age: 3-65 years
* Measurable overgrowth, in current progression or with clinical history of overgrowth progression
* Patient clinically stable
* Presence of a disability, social or cosmetic impairment requiring treatment from the patient perspective,
* Written informed consent form signed and dated by the subject or by the patient's legal representative

Exclusion Criteria:

* Pregnancy or lactation
* Women and men of reproductive age without any effective method of contraception (during treatment and up to 12 weeks after sirolimus discontinuation)
* Hypersensitivity to the active substance (sirolimus) or to any of the excipients
* Impossibility to obtain written informed consent form signed by the subject or the patient's legal representative, or vulnerable adults
* Treatment with Sirolimus in the last 4 weeks before the trial
* Personal history of malignancy or current investigations for suspected malignancy
* Active skin infection requiring antibiotics or antiviral treatments
* HIV or hepatitis B or C infection
* Past history of Mycobacterium tuberculosis infection
* Active pneumopathy
* Uncontrolled infection
* Chronic liver disease (ASAT or Alanine amino transférase (ALAT)> 3 times upper normal limit)
* Stage 3 (or more) chronic renal insufficiency (eGFR< 60mls/min)
* Neutropenia with neutrophiles < 1.0 x10^9/L
* Uncontrolled dyslipidemia
* Inability to attend study visits

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measure of the relative percentage of the excess tissue volume evolution at the affected site by volumetric MRI. | Change from baseline at 6 and 12 months

SECONDARY OUTCOMES:
Measure sites of overgrowth by DXA, MRI and circumferential measurements | Change from baseline at 6 and 12 months
To determine optimal sirolimus dosing algorithms by plasma assay | 12 months
Number of hospitalisation and surgery | 12 months
quality of life measured by a questionnaire in the pre- and post-treatment periods | At 6 and 12 months
  The WHO-QOL-BREF questionnaire will be used for adults. For children, PedsQL™ questionnaire for children and parents report for children questionnaires will be used

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHU de Bordeaux - GH Pellegrin, Bordeaux
  - CHU de DIJON, Dijon
  - Hôpital Jeanne de Flandre, Lille
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - Hopitaux de Brabois Chu Nancy, Nancy
  - Hôpital mère-enfant de Nantes, Nantes
  - CHU Paris - Necker, Paris
  - HCL Lyon - CH Lyon Sud, Pierre-Bénite
  - Pôle Cardiovasculaire et Métabolique - Hôpital Larrey, Toulouse
  - CHRU de Tours, Tours

REFERENCES:
- [Result] Parker VER, Keppler-Noreuil KM, Faivre L, Luu M, Oden NL, De Silva L, Sapp JC, Andrews K, Bardou M, Chen KY, Darling TN, Gautier E, Goldspiel BR, Hadj-Rabia S, Harris J, Kounidas G, Kumar P, Lindhurst MJ, Loffroy R, Martin L, Phan A, Rother KI, Widemann BC, Wolters PL, Coubes C, Pinson L, Willems M, Vincent-Delorme C; PROMISE Working Group; Vabres P, Semple RK, Biesecker LG. Safety and efficacy of low-dose sirolimus in the PIK3CA-related overgrowth spectrum. Genet Med. 2019 May;21(5):1189-1198. doi: 10.1038/s41436-018-0297-9. Epub 2018 Oct 1. PMID 30270358